CLINICAL TRIAL: NCT02666937
Title: Safe Limits in Saturation (SLIM-study)
Acronym: SLIM
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Angelique Spoelstra-de Man, Dr. A.M.E. Spoelstra--de Man, Amsterdam UMC, location VUmc
Other Study IDs: 2014.524 (A2015.361)
Record Dates: First submitted 2015-11-30; First posted 2016-01-28 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Critical Illness; Hyperoxia; Hypoxia
MeSH Terms: conditions — Critical Illness; Hyperoxia; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- ICU-patients (prospective): Critically ill patients (18 years and older) on mechanically ventilation who have an arterial line and require bloodgasanalysis for medical reasons
- Emergency Department (prospective): Patients (18 years and older), who are presented to the Emergency Department, and require bloodgasanalysis for medical reasons
- Pulmonary department (prospective): Patients (18 years and older) who visit the outpatient clinic of the pulmonary department for different pulmonary functional test and require bloodgasanalysis for medical reasons
- Pulmonary department (retrospective): Patients (18 years and older) who visited the outpatient clinic of the pulmonary department in the past of the VU medical centre in Amsterdam or the Medical Centre Alkmaar for different pulmonary functional test and required bloodgasanalysis for medical reasons

SUMMARY:
A study consisting of a prospective and retrospective cohort in the ICU, ER and pulmonary department in a university hospital in Amsterdam and a teaching hospital in Alkmaar, the Netherlands.

The relationship between the oxygen saturation measured by pulse-oximetry and the arterial PaO2 is investigated in order to investigate which transcutaneous saturation values are safe when administering oxygen in relation to hyperopia and hypoxia.

DETAILED DESCRIPTION:
This study consists of two parts a prospective and a retrospective part.

1. Prospective part: Patients in the ICU, the emergency room and the pulmonary function department of the VU university medical centre will be included. Arterial blood gas analysis is a tool often used to determine PaO2 in regular care. When an arterial blood gas analysis is performed for regular patient care, the corresponding SpO2 is measured. Information such as blood pressure, heart rate, amount of administered fluids and shock-related-parameters are obtained from the patient files. For the ICU patients capillary refill, acra temperature and the mottling scores are examined. The peripheral flow index and temperature index is measured. When more arterial blood gas samples are drawn over time in one patient, multiple datasets can be included per patient, as long as the samples are drawn two hours apart.
2. Retrospective part: Patients with a (suspected) pulmonary disease who underwent pulmonary function tests with arterial bloodgas sampling in the VU medical center and Medical Centre Alkmaar in the last 25 years. The PaO2 and corresponding SpO2 will be obtained from the test and parameters such as blood pressure, heart rate and administered oxygen will be retrieved from the databases with these test results.

ELIGIBILITY:
Inclusion criteria for all inclusions:

* Age: 18>
* Requiring arterial bloodgas analysis

Exclusion criteria for all inclusions:

* Hyperbilirubinemia (>20 μmol/L)
* CO-Hb (>1,5%)
* MetHb (>1,5%)
* Unreliable pulsatile SpO2 curve

Additional inclusion criteria:

- Prospective, ICU - VUmc: On mechanical ventilation. Arterial line in place.

Additional exclusion criteria:

* Prospective, ICU - VUmc: On extracorporeal membrane oxygenation. Therapeutic hypothermia.
* Retrospective, Pulmonary function departments: Uncertainty whether SpO2 was measured exactly during arterial bloodgas sampling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective
  * ICU - VUmc: Critically ill patients, requiring invasive monitoring
  * Pulmonary function department - VUmc: Patients requiring a pulmonary function test with arterial bloodgas analysis.
  * ER VUmc: Patients presented at the shockroom or patients in the general ER, requiring arterial bloodgas analysis.
  Retrospective
  - Pulmonary function departments: Patients who underwent a pulmonary function test with arterial bloodgas analysis in the last 25 years.
Sampling Method: Probability Sample
Enrollment: 879 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Relation SpO2-PaO2 | Average of one week
  To determine peripherally measured saturation targets between which no hyperoxia and hypoxia will occur

SECONDARY OUTCOMES:
Factors influencing PaO2-Spo2 relation | Average of one week
  To identify factors influencing the relationship between SpO2 and PaO2, such as hemodynamics, peripheral circulation, shock and pH
Relation in SpO2-PaO2 in different populations | Average of one week
  To determine differences in the SpO2/PaO2 -relationship in different populations
Differences in relation in SpO2-PaO2 prospective versus retrospective | Average of one week
  To determine differences in the SpO2/PaO2 -relationship in a prospective and a retrospective cohort

CONTACTS AND LOCATIONS:
Overall Officials: Angelique ME Spoelstra - de Man, Phd Md, Study Director — Amsterdam UMC, location VUmc
Locations (1):
- VUMedicalCentre, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Background] Cornet AD, Kooter AJ, Peters MJ, Smulders YM. Supplemental oxygen therapy in medical emergencies: more harm than benefit? Arch Intern Med. 2012 Feb 13;172(3):289-90. doi: 10.1001/archinternmed.2011.624. Epub 2012 Jan 9. No abstract available. PMID 22231614
- [Background] de Jonge E, Peelen L, Keijzers PJ, Joore H, de Lange D, van der Voort PH, Bosman RJ, de Waal RA, Wesselink R, de Keizer NF. Association between administered oxygen, arterial partial oxygen pressure and mortality in mechanically ventilated intensive care unit patients. Crit Care. 2008;12(6):R156. doi: 10.1186/cc7150. Epub 2008 Dec 10. PMID 19077208
- [Background] Austin MA, Wills KE, Blizzard L, Walters EH, Wood-Baker R. Effect of high flow oxygen on mortality in chronic obstructive pulmonary disease patients in prehospital setting: randomised controlled trial. BMJ. 2010 Oct 18;341:c5462. doi: 10.1136/bmj.c5462. PMID 20959284
- [Background] Kilgannon JH, Jones AE, Shapiro NI, Angelos MG, Milcarek B, Hunter K, Parrillo JE, Trzeciak S; Emergency Medicine Shock Research Network (EMShockNet) Investigators. Association between arterial hyperoxia following resuscitation from cardiac arrest and in-hospital mortality. JAMA. 2010 Jun 2;303(21):2165-71. doi: 10.1001/jama.2010.707. PMID 20516417
- [Background] Kuisma M, Boyd J, Voipio V, Alaspaa A, Roine RO, Rosenberg P. Comparison of 30 and the 100% inspired oxygen concentrations during early post-resuscitation period: a randomised controlled pilot study. Resuscitation. 2006 May;69(2):199-206. doi: 10.1016/j.resuscitation.2005.08.010. Epub 2006 Feb 24. PMID 16500018
- [Background] Bellomo R, Bailey M, Eastwood GM, Nichol A, Pilcher D, Hart GK, Reade MC, Egi M, Cooper DJ; Study of Oxygen in Critical Care (SOCC) Group. Arterial hyperoxia and in-hospital mortality after resuscitation from cardiac arrest. Crit Care. 2011;15(2):R90. doi: 10.1186/cc10090. Epub 2011 Mar 8. PMID 21385416
- [Background] Meyhoff CS, Jorgensen LN, Wetterslev J, Christensen KB, Rasmussen LS; PROXI Trial Group. Increased long-term mortality after a high perioperative inspiratory oxygen fraction during abdominal surgery: follow-up of a randomized clinical trial. Anesth Analg. 2012 Oct;115(4):849-54. doi: 10.1213/ANE.0b013e3182652a51. Epub 2012 Jul 13. PMID 22798533
- [Background] Quintard H, Patet C, Suys T, Marques-Vidal P, Oddo M. Normobaric hyperoxia is associated with increased cerebral excitotoxicity after severe traumatic brain injury. Neurocrit Care. 2015 Apr;22(2):243-50. doi: 10.1007/s12028-014-0062-0. PMID 25168744
- [Background] Rincon F, Kang J, Maltenfort M, Vibbert M, Urtecho J, Athar MK, Jallo J, Pineda CC, Tzeng D, McBride W, Bell R. Association between hyperoxia and mortality after stroke: a multicenter cohort study. Crit Care Med. 2014 Feb;42(2):387-96. doi: 10.1097/CCM.0b013e3182a27732. PMID 24164953
- [Background] Baleeiro CE, Wilcoxen SE, Morris SB, Standiford TJ, Paine R 3rd. Sublethal hyperoxia impairs pulmonary innate immunity. J Immunol. 2003 Jul 15;171(2):955-63. doi: 10.4049/jimmunol.171.2.955. PMID 12847267
- [Background] Davis WB, Rennard SI, Bitterman PB, Crystal RG. Pulmonary oxygen toxicity. Early reversible changes in human alveolar structures induced by hyperoxia. N Engl J Med. 1983 Oct 13;309(15):878-83. doi: 10.1056/NEJM198310133091502. PMID 6888481
- [Background] Jackson RM. Pulmonary oxygen toxicity. Chest. 1985 Dec;88(6):900-5. doi: 10.1378/chest.88.6.900. PMID 3905287
- [Background] Fracica PJ, Knapp MJ, Piantadosi CA, Takeda K, Fulkerson WJ, Coleman RE, Wolfe WG, Crapo JD. Responses of baboons to prolonged hyperoxia: physiology and qualitative pathology. J Appl Physiol (1985). 1991 Dec;71(6):2352-62. doi: 10.1152/jappl.1991.71.6.2352. PMID 1778933
- [Background] Harten JM, Anderson KJ, Angerson WJ, Booth MG, Kinsella J. The effect of normobaric hyperoxia on cardiac index in healthy awake volunteers. Anaesthesia. 2003 Sep;58(9):885-8. doi: 10.1046/j.1365-2044.2003.03333.x. PMID 12911363
- [Background] Lodato RF. Decreased O2 consumption and cardiac output during normobaric hyperoxia in conscious dogs. J Appl Physiol (1985). 1989 Oct;67(4):1551-9. doi: 10.1152/jappl.1989.67.4.1551. PMID 2793757
- [Background] Haque WA, Boehmer J, Clemson BS, Leuenberger UA, Silber DH, Sinoway LI. Hemodynamic effects of supplemental oxygen administration in congestive heart failure. J Am Coll Cardiol. 1996 Feb;27(2):353-7. doi: 10.1016/0735-1097(95)00474-2. PMID 8557905
- [Background] Zwemer CF, Whitesall SE, D'Alecy LG. Cardiopulmonary-cerebral resuscitation with 100% oxygen exacerbates neurological dysfunction following nine minutes of normothermic cardiac arrest in dogs. Resuscitation. 1994 Mar;27(2):159-70. doi: 10.1016/0300-9572(94)90009-4. PMID 8086011
- [Background] O'Driscoll BR, Howard LS, Davison AG; British Thoracic Society. BTS guideline for emergency oxygen use in adult patients. Thorax. 2008 Oct;63 Suppl 6:vi1-68. doi: 10.1136/thx.2008.102947. No abstract available. PMID 18838559
- [Background] Decalmer S, O'Driscoll BR. Oxygen: friend or foe in peri-operative care? Anaesthesia. 2013 Jan;68(1):8-12. doi: 10.1111/anae.12088. Epub 2012 Nov 7. No abstract available. PMID 23130783
- [Background] Suzuki S, Eastwood GM, Glassford NJ, Peck L, Young H, Garcia-Alvarez M, Schneider AG, Bellomo R. Conservative oxygen therapy in mechanically ventilated patients: a pilot before-and-after trial. Crit Care Med. 2014 Jun;42(6):1414-22. doi: 10.1097/CCM.0000000000000219. PMID 24561566
- [Background] Sinex JE. Pulse oximetry: principles and limitations. Am J Emerg Med. 1999 Jan;17(1):59-67. doi: 10.1016/s0735-6757(99)90019-0. PMID 9928703
- [Background] Nitzan M, Romem A, Koppel R. Pulse oximetry: fundamentals and technology update. Med Devices (Auckl). 2014 Jul 8;7:231-9. doi: 10.2147/MDER.S47319. eCollection 2014. PMID 25031547
- [Background] Swain DP, Pittman RN. Oxygen exchange in the microcirculation of hamster retractor muscle. Am J Physiol. 1989 Jan;256(1 Pt 2):H247-55. doi: 10.1152/ajpheart.1989.256.1.H247. PMID 2912188
- [Background] Jensen LA, Onyskiw JE, Prasad NG. Meta-analysis of arterial oxygen saturation monitoring by pulse oximetry in adults. Heart Lung. 1998 Nov-Dec;27(6):387-408. doi: 10.1016/s0147-9563(98)90086-3. PMID 9835670
- [Background] Astiz ME, Rackow EC, Kaufman B, Falk JL, Weil MH. Relationship of oxygen delivery and mixed venous oxygenation to lactic acidosis in patients with sepsis and acute myocardial infarction. Crit Care Med. 1988 Jul;16(7):655-8. doi: 10.1097/00003246-198807000-00001. PMID 3371040
- [Background] van Genderen ME, Lima A, Bakker J, van Bommel J. [Peripheral circulation in critically ill patients: non-invasive methods for the assessment of the peripheral perfusion]. Ned Tijdschr Geneeskd. 2013;157(9):A5338. Dutch. PMID 23446154
- [Background] House JR, Tipton MJ. Using skin temperature gradients or skin heat flux measurements to determine thresholds of vasoconstriction and vasodilatation. Eur J Appl Physiol. 2002 Nov;88(1-2):141-5. doi: 10.1007/s00421-002-0692-3. Epub 2002 Sep 3. PMID 12436282
- [Background] Sessler DI. Skin-temperature gradients are a validated measure of fingertip perfusion. Eur J Appl Physiol. 2003 May;89(3-4):401-2; author reply 403-4. doi: 10.1007/s00421-003-0812-8. Epub 2003 Mar 25. No abstract available. PMID 12736848
- [Background] Durlinger EMJ, Spoelstra-de Man AME, Smit B, de Grooth HJ, Girbes ARJ, Oudemans-van Straaten HM, Smulders YM. Hyperoxia: At what level of SpO2 is a patient safe? A study in mechanically ventilated ICU patients. J Crit Care. 2017 Jun;39:199-204. doi: 10.1016/j.jcrc.2017.02.031. Epub 2017 Mar 2. PMID 28279497